CLINICAL TRIAL: NCT01186484
Title: Phase 1 Study of JNJ-212082 (Abiraterone Acetate) in Patients With Castration-Resistant Prostate Cancer
Brief Title: Phase 1 Study of Abiraterone Acetate in Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017137; JNJ-212082-JPN-102 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Neoplasms
Keywords: Castration-resistant prostate cancer; Abiraterone acetate; JNJ-212082
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- 001 (Experimental): JNJ-212082 250 mg 500 mg or 1000 mg once daily up to discontinuation for any reasons such as progression of the disease or up to the transition to extension study.
  Interventions: Drug: JNJ-212082

INTERVENTIONS:
Drug: JNJ-212082 — 250 mg, 500 mg or 1000 mg once daily up to discontinuation for any reasons such as progression of the disease or up to the transition to extension study.

SUMMARY:
The purpose of this study is to assess pharmacodynamics and safety of JNJ-212082 in order to select the recommended dose of JNJ-212082 for patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
This study is a multicenter (more than one site), open-label (both physician and patient know the name of the study drug), dose-escalation study in chemotherapy-naive patients with castration- resistant prostate cancer (CRPC) to evaluate the pharmacodynamics (the study of the action or effects of drugs on living organisms), safety, pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) and preliminary effectiveness of JNJ-212082. The dose of the study will be escalated from 250 mg (cohort 1), 500 mg (cohort 2), to 1000 mg (cohort 3). Six to twelve patients within each 250 mg, 500 mg or 1000 mg cohort will be orally administered drug once per day. Comprising 28 days for each 1 cycle, the administration will be continued up to discontinuation for any reasons such as progression of the disease or up to the transition to extension study (Protocol number: JNJ-212082-JPN-203) which will be separately planned. In addition, 5 mg of prednisolone will be orally administered twice per day since Day 8. On receiving notification of the confirmation of safety of 500 mg of the drug, patients of cohort 1 who are currently on continuous administration can receive increment 500 mg per day starting from the next cycle (If the dose escalation would not be appropriate due to safety reasons, the patients will continue the original dose). Furthermore, on receiving notification of the confirmation of safety of 1000 mg, patients of previous cohorts who are currently on continuous administration can receive increment 1000 mg per day as well from the next cycles (If the dose escalation would not be appropriate due to safety reasons, the patients will continue the original dose). JNJ-212082 will be orally administered once per day. Comprising 28 days for each 1 cycle, the administration will be continued up to discontinuation for any reasons such as progression of the disease or up to the transition to extension study. The drug will be administered at least 1 hour prior to meal or 2 hours after meal. The daily dose of the drug is defined as 250 mg, 500 mg or 1000 mg. In addition, 5 mg of prednisolone (marketed) will be orally administered twice per day since Day 8.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate, but not with neuroendocrine differentiation or of small cell histology
* No Prior cytotoxic chemotherapy (including estramustine) for the treatment of prostate cancer
* Surgically or medically castrated, with testosterone levels of < 0.5 ng/mL
* PSA level of at least 2 ng/ml at Screening
* PSA progression according to PCWG2 eligibility criteria or objective progression by RECIST criteria for patients with measurable disease after androgen deprivation

Exclusion Criteria:

* Surgery or local prostatic intervention within 4 weeks of the first dose. In addition, any clinically relevant sequelae from the surgery have not resolved prior to initial treatment
* Radiotherapy, or immunotherapy within 4 weeks, or single fraction of palliative radiotherapy within 2 weeks of administration prior to initial treatment
* Known brain metastasis
* Uncontrolled hypertension (systolic BP greater than 160 mmHg or diastolic BP greater than 95 mmHg)
* Active or symptomatic viral hepatitis or chronic liver disease

Ages: 20 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2014-10-02 (Actual); Study Completion 2014-10-02 (Actual)

PRIMARY OUTCOMES:
The pharmacodynamics (serum concentrations of corticosterone, testosterone, DHEA-S, 11-deoxycorticosterone) | At Days 1, 2, and 8 of Cycle 1
The number of patients reporting adverse events as a measure of safety | 4 weeks

SECONDARY OUTCOMES:
Plasma concentrations of abiraterone acetate and abiraterone | 4 weeks
Rates of decrease of prostate specific antigen (PSA)>50% (criteria of PCWG2 - Prostate Cancer Clinical Trials Working Group) | Maximum 52 weeks
Tumor regression in patients with measurable lesions (RECIST - Response evaluation criteria in solid tumors) | Maximum 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - Fukuoka
  - Kashiwa
  - Kōtoku
  - Sunto
  - Yokohama

REFERENCES:
- [Derived] Matsubara N, Uemura H, Fukui I, Niwakawa M, Yamaguchi A, Iizuka K, Akaza H. Phase-1 study of abiraterone acetate in chemotherapy-naive Japanese patients with castration-resistant prostate cancer. Cancer Sci. 2014 Oct;105(10):1313-20. doi: 10.1111/cas.12496. Epub 2014 Oct 4. PMID 25117615
- See also: Phase 1 study of JNJ-212082 (abiraterone acetate) in Chemotherapy-Naïve Patients With Castration-Resistant Prostate Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=438&filename=JNJ-212082-JPN-102-Synopsis.pdf